CLINICAL TRIAL: NCT07205094
Title: Effect of Telerehabilitation Versus Conventional Physiotherapy on Quality of Life, Pain, and Functional Outcomes in Patients Following Rotator Cuff Surgery
Brief Title: Effect of Telerehabilitation on Quality of Life, Pain, and Function After Rotator Cuff Surgery
Acronym: TELERO-ROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysan Yaghoubi (Other)
Responsible Party: Sponsor-Investigator, Aysan Yaghoubi, Master's Graduate in Physiotherapy and Rehabilitation, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AYSAN2025-RCT
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Surgery; Telerehabilitation Method; Pain; Quality of Life; Function
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Intervention Model Description: Participants were assigned to two groups: a telerehabilitation group (n=20) and a conventional physiotherapy control group (n=10). Both groups followed an eight-week exercise program, including range of motion, stretching, strengthening, and stabilization exercises. Outcomes such as pain, shoulder mobility, muscle strength, functional ability, and quality of life were compared between the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): 8-week telerehabilitation program including range of motion, stretching, strengthening, and stabilization exercises
  Interventions: Other: Telerehabilitation exercise program
- Conventional Physiotherapy (Active Comparator): 8-week conventional face-to-face physiotherapy program including range of motion, stretching, strengthening, and stabilization exercises
  Interventions: Other: Conventional physiotherapy program

INTERVENTIONS:
Other: Telerehabilitation exercise program — 8-week telerehabilitation program including range of motion, stretching, strengthening, and stabilization exercise
  Arms: Telerehabilitation
Other: Conventional physiotherapy program — 8-week conventional face-to-face physiotherapy program including range of motion, stretching, strengthening, and stabilization exercises
  Arms: Conventional Physiotherapy

SUMMARY:
he purpose of this study was to find out whether telerehabilitation after rotator cuff surgery can help reduce pain, improve shoulder movement, increase muscle strength, enhance functional ability, and improve quality of life compared to conventional physiotherapy. The study included 30 participants who had undergone rotator cuff surgery at least six weeks earlier. They were divided into two groups: a telerehabilitation group (n=20) and a conventional physiotherapy control group (n=10). Both groups followed an eight-week exercise program, which included range of motion, stretching, strengthening, and stabilization exercises.

The study found that both groups improved in pain, shoulder mobility, muscle strength, function, and quality of life. Participants in the telerehabilitation group showed particularly greater improvements in shoulder flexion, flexor muscles, external rotator muscles, and overall quality of life. These results suggest that telerehabilitation may be an effective alternative to traditional physiotherapy after rotator cuff surgery.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone rotator cuff surgery
* At least 6 weeks post-surgery
* Possess the necessary technology for telerehabilitation (smartphone, computer, internet access)
* Willing to participate in the study and have signed the informed consent form

Exclusion Criteria:

* History of neurological disorders
* Severe cardiovascular or pulmonary conditions
* Need for special medical care due to postoperative infection or complications
* Inability to comply with telerehabilitation due to psychiatric conditions
* Lack of access to or knowledge of technology required for telerehabilitation
* Participation in another rehabilitation program during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity (Visual Analog Scale [VAS], 0-10 points) | Baseline and after 8-week intervention
  Pain intensity was assessed before and after the 8-week intervention using the Visual Analog Scale (VAS) during activity, at rest, and at night. Scores range from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating worse pain. Changes were compared between the telerehabilitation group and the conventional physiotherapy control group.

SECONDARY OUTCOMES:
Shoulder range of motion (Goniometer, degrees) | Baseline and after 8-week intervention
  Shoulder flexion, extension, abduction, adduction, internal rotation, and external rotation were measured using a goniometer before and after the 8-week intervention. Normal ranges for adults are: flexion 0-180°, extension 0-45°, abduction 0-180°, adduction 0-45°, internal rotation 0-70°, external rotation 0-90°. Changes were compared between the telerehabilitation group and control group.
Muscle strength (Manual Muscle Testing, 0-5 scale) | Baseline and after 8-week intervention
  Muscle strength of shoulder flexors, extensors, abductors, adductors, internal and external rotators was assessed using manual muscle testing before and after the 8-week intervention. Scores range from 0 (no contraction) to 5 (normal strength), with higher scores indicating stronger muscles. Changes were compared between groups.
Quality of life (Western Ontario Rotator Cuff Index [WORC], 0-2100 points) | Baseline and after 8-week intervention
  Quality of life was assessed before and after the 8-week intervention using the WORC questionnaire. Scores range from 0 (best quality of life) to 2100 (worst quality of life), with lower scores indicating better quality of life. Changes were compared between the telerehabilitation group and control group.
Functional status (Disabilities of the Arm, Shoulder, and Hand [DASH] questionnaire, 0-100 points) | Baseline and after 8-week intervention.
  Functional status was measured before and after the 8-week intervention using the DASH questionnaire. Scores for each subscale (function, symptoms, social/role function) were calculated separately. Scores range from 0 (no disability) to 100 (maximum disability), with higher scores indicating worse functional status. Changes were compared between the telerehabilitation group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Beykent University Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT07205094/ICF_000.pdf